CLINICAL TRIAL: NCT04585906
Title: My Pathway to Healing: Adaptation and Testing of a Common Elements Treatment Approach to Address Trauma, Suicide Ideation and Substance Abuse
Brief Title: My Pathway to Healing
Acronym: MP2H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Native American Research Center for Health (Other); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JHSPH-9500; 1S06GM127981 (NIH); IRB00009500 (Other: JHSPH IRB)
Record Dates: First submitted 2020-08-26; First posted 2020-10-14 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Suicide; Trauma; Binge Drinking
MeSH Terms: conditions — Suicide; Wounds and Injuries; Binge Drinking

STUDY DESIGN:
Intervention Model Description: Investigators will use a randomized control design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sessions with a community mental health specialist (Experimental): Those randomized into the intervention group will receive 4-8 hour-long sessions with a community mental health specialist, taking place over approximately 12 weeks. The common elements treatment approach intervention (called "My Pathway to Healing") includes psychoeducation and addresses safety (when identified as a problem area). It also includes relaxation techniques, problem solving, and cognitive coping. The exact number of sessions delivered will depend on presentation and symptom level using a stepped care approach where participants receive only what they need, but the provider can provide additional sessions if needed (i.e., increased element dosage; additional optional elements for specific issues).
  Interventions: Behavioral: Common Elements Treatment Approach
- Case management (Active Comparator): This study employs a randomized control design in which participants in the control group will receive case management and offered the intervention upon completion of their enrollment period.
  Interventions: Behavioral: Common Elements Treatment Approach

INTERVENTIONS:
Behavioral: Common Elements Treatment Approach — The intervention integrates psychoeducation and addresses safety (when identified as a problem area). It also includes relaxation techniques, problem solving, and cognitive coping.

SUMMARY:
The goal of this project is to test the feasibility and acceptability of a common elements intervention delivered by community mental health workers for adults with a history of adverse childhood experiences. "Common elements" interventions build cognitive, emotional, interpersonal, and behavioral skills to help address trauma-related distress and build resilience. This will be accomplished using a randomized control trial with Apache adults ages 25-65 with recent suicidal behaviors, self-injurious behaviors, and/or binge substance use.

DETAILED DESCRIPTION:
This is a mixed-methods study with qualitative data informing adaptation and evaluation of a common elements intervention delivered by community mental health specialists, named "My Pathway to Healing." The study includes a pilot trial and CAB discussions to inform our understanding of the feasibility of scaling up the intervention.

The investigators randomized some participants to receive the interventions and some to receive control case manager visits, to pilot what a future effectiveness RCT might be. This intervention integrates psychoeducation, relaxation techniques, problem solving and cognitive coping, and addresses safety (when identified as a problem area). The intervention used in the intervention arm of our study has been developed for the specific context and culture of White Mountain Apache.

Those randomized into the My Pathway to Healing group will receive 4-8 hour-long sessions with a community mental health specialist, taking place over 8-12 weeks. The exact number of sessions will depend on presentation and symptom level using a stepped care approach where participants receive only what they need, but the provider can provide additional sessions if needed (i.e., increased element dosage; additional optional elements for specific issues). Those randomized into the control will continue to receive the standard case management via the Apache surveillance system. These control participants will be offered the My Pathway to Healing Program upon completion of the study.

Participants will be asked to partake in 5 study assessments. For intervention participants these assessments will take place at: baseline, after their last intervention session (endline; approximately 8-12 weeks post-baseline) and 4, 8, and 12 weeks post-endline. For control participants, these assessments will take place at: baseline, 8-12 weeks post-baseline (the maximum time the intervention would last; will be referred to as an endline) and 4, 8 and 12 weeks post-endline. These assessment visits will be conducted by Research Program Assistants. Assessments will take approximately 45-90 minutes to complete. In the feasibility study, assessments are not being statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 25-65
* Suicide ideation, suicide attempt, self-injurious behavior, and/or binge alcohol and/or drug use within past 90 days confirmed by the Apache suicide surveillance system
* Experienced at least 2 adverse childhood experiences
* Native American
* Reside on or near the Fort Apache Indian Reservation.
* An average score of 1 or above on a measure of symptoms of posttraumatic stress

Exclusion Criteria:

* Unable to provide informed consent
* Have a serious developmental disorder
* Have active psychosis

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Haroz, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Center for American Indian Health Whiteriver Office, Whiteriver, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Data collected as part of this project is protected by tribal sovereignty. Any requests for data sharing must be approved by all relevant tribal authorities (tribal council, health board, etc.) before data can be shared.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consented n=36 adults, then n=5 were lost to followup (LTFU) before baseline assessment; n=31 completed baseline assessment and were randomized.
Period: Overall Study
Arm/Group | Sessions With a Community Mental Health Specialist | Case Management
Started | 15 | 16
Completed | 7 | 11
Not Completed | 8 | 5
Not completed — Lost to Follow-up | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sessions With a Community Mental Health Specialist | Case Management | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 16 | 31
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 8 | 12 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 15 | 16 | 31
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 16 | 31
Index event behavior [Count of Participants; unit: Participants] — Participants were eligible for the study with self-injury, binge substance use, suicide ideation or attempt.
  Participants
    Binge substance use | 5 | 8 | 13
    Self-injury | 1 | 1 | 2
    Suicide ideation | 7 | 6 | 13
    Suicide attempt | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Completing Visits
Description: Feasibility as assessed by the number of participants completing sessions; 0, 0% reflects lowest feasibility, 100% reflects highest feasibility.
Time Frame: Up to 12 weeks post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Sessions With a Community Mental Health Specialist | Case Management
Number analyzed (Participants) | 15 | 16
Participants | 7 | 11

2. Primary Outcome: Number of People Approached Who Consented or Declined
Description: This timepoint is pre-randomization. 68 potential participants were approached to join the study; feasible if those who decline participation is less than 20%, a lower decline percentage indicates greater feasibility. A higher consent percentage indicates greater feasibility.
Time Frame: At consent
Population: Potential participants approached
Measure: Count of Participants; unit: Participants
Groups:
- Declined: Potential participants were deemed eligible for study participation, approached for consent, and declined participation.
- Consented: Potential participants were deemed eligible for study participation, approached for consent, and consented to participation.
Arm/Group | Declined | Consented
Number analyzed (Participants) | 68 | 68
Participants | 32 | 36

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Sessions With a Community Mental Health Specialist | Case Management
All-Cause Mortality (participants affected / at risk) | 1/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 1/15 | 2/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sessions With a Community Mental Health Specialist (N=15) | Case Management (N=16)
Binge substance use (Social circumstances) | 0 (0) | 2 (11) — Participant had binge substance use reported
Suicide ideation (Psychiatric disorders) | 1 (1) | 0 (0) — Suicide ideation reported

LIMITATIONS AND CAVEATS:
Investigators received sponsor approval to transition the randomized control trial to a feasibility study with smaller sample size. Investigators aimed to recruit 30 participants and understand the feasibility of scaling this study at a larger size and understand the challenges of implementing this intervention with this population of adults experiencing suicide, self-injury, and substance use. The rest of the study design, aside from the sample size, remained the same throughout the project.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-27): https://cdn.clinicaltrials.gov/large-docs/06/NCT04585906/Prot_SAP_003.pdf
  • Informed Consent Form (2022-05-27): https://cdn.clinicaltrials.gov/large-docs/06/NCT04585906/ICF_004.pdf